CLINICAL TRIAL: NCT06066489
Title: Effect of Educational Program for Nurses About Preventive Care Bundle for Prevention of Ventilator Associated Pneumonia Among Newborns
Brief Title: Effect of Educational Program About Preventive Care Bundle for Prevention of Ventilator Associated Pneumonia Among Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Basma Ibrahim, lecturer, Damanhour University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VAP in newborns
Record Dates: First submitted 2023-09-22; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Ventilator Associated Pneumonia
Keywords: newborn
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: A prospective, quasi-experimental, pre- and post-study with a one month baseline period; one month intervention period and three months post-intervention period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurses (Experimental): Nurses will be assessed first about their knowledge about VAP then they will receive an educational program about VAP and will be assessed immediately and 3 months after the program
  Interventions: Other: educational program about VAP
- newborns (Experimental): the prevalence of VAP will be assessed among all ventilated newborns who will meet inclusion criteria in the study before implementing the program, immediately and 3 months after the program using PNU1
  Interventions: Other: educational program about VAP

INTERVENTIONS:
Other: educational program about VAP — An educational program about VAP that includes VAP bundle from CDC as core measures , equipment related measures and general measures.

SUMMARY:
This study is designed to investigate the effect of educational program for nurses about preventive care bundle for prevention of ventilator associated pneumonia among newborns.

DETAILED DESCRIPTION:
Neonatal ventilator associated pneumonia (VAP) is a common nosocomial infection and a frequent reason for empirical antibiotic therapy in NICUs. Ventilator associated pneumonia (VAP) is defined as a nosocomial lower airway infection in intubated patients with onset after 48 h or more of invasive mechanical ventilation.Prevention of VAP has been primarily achieved by the "bundle approach"; this involves the simultaneous application of several preventive strategies for all patients.In Egypt and other developing countries, reports on the success of VAP intervention strategies, particularly among neonates, are scarce. So, it is important to conduct educational programs for nurses about VAP to decrease its incidence.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥34 weeks
* Intubated newborns and those expected to receive mechanical ventilation for more than 48 hours.

Exclusion Criteria:

* Newborns with diagnosis of pneumonia at the time of admission.
* Newborns developed pneumonia in the first 48 hours of mechanical ventilation.
* Newborns subjected to reintubation.
* Immunosuppressed newborns.

Ages: 3 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
prevalence of VAP among newborns ( the number of newborns diagnosed with VAP during the study period | before intervention as baseline ( Day 1), immediately after the intervention, 3 months later after intervention
  prevalence of VAP will be compared before application of educational program for nurses about preventive care bundle for prevention of VAP and after the program ( immediately, 3 months later) by using centers for disease control and prevention PNU-1

SECONDARY OUTCOMES:
nurses practices about prevention of ventilator associated pneumonia after implementing the training program will be compared by their practices before the intervention using Observational Checklist | before intervention as baseline(Day 1), immediately after the intervention, 3 months later after intervention
  nurses practices will be assessed before and after the intervention immediately and 3 months later using Observational Checklist about their practices and then results compared before and after the intervention by mean percent score

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iosifidis E, Pitsava G, Roilides E. Ventilator-associated pneumonia in neonates and children: a systematic analysis of diagnostic methods and prevention. Future Microbiol. 2018 Sep;13:1431-1446. doi: 10.2217/fmb-2018-0108. Epub 2018 Sep 26. PMID 30256161
- [Background] Alriyami A, Kiger JR, Hooven TA. Ventilator-Associated Pneumonia in the Neonatal Intensive Care Unit. Neoreviews. 2022 Jul 1;23(7):e448-e461. doi: 10.1542/neo.23-7-e448. PMID 35773508
- [Background] Niedzwiecka T, Patton D, Walsh S, Moore Z, O'Connor T, Nugent L. What are the effects of care bundles on the incidence of ventilator-associated pneumonia in paediatric and neonatal intensive care units? A systematic review. J Spec Pediatr Nurs. 2019 Oct;24(4):e12264. doi: 10.1111/jspn.12264. Epub 2019 Jul 23. PMID 31332968